CLINICAL TRIAL: NCT00248274
Title: Assessment of Atrial Tissue Obtained From Patients Undergoing Heart Surgery
Brief Title: Atrial Tissue Banking: Atrial Tissue Obtained From Patients Undergoing Heart Surgery
Status: Terminated | Type: Observational
Why Stopped: Staffing and departmental changes at our site made it difficult to enroll subjects.
Sponsor: University of Pittsburgh (Other)
Collaborators: EP Research funds (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0406094
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; genetics
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. myocardial tissue
  2. DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Over the past decade, techniques have been refined which permit an enormous amount of information relevant to disease mechanisms to be gained from the examination of heart tissue. The Cardiovascular Institute has extensive experience with these techniques, and has utilized them to examine other heart disease substrates.

In this study, the investigators propose to obtain heart tissue at the time of cardiac surgery which would otherwise be discarded. Their plan is to examine this tissue and correlate their findings with clinical data. Their hope is that the proposed study will provide insight into atrial physiology, including the molecular mechanisms underlying atrial disease and the potential development of atrial fibrillation (AF).

This will be a prospective "registry" for atrial tissue. The investigators propose an enrollment of 300 subjects, to take place at University of Pittsburgh Medical Center (UPMC) Presbyterian over a 5 year period.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), a disorder of heart rhythm, is epidemic in the United States, affecting nearly 3 million people. AF arises in a variety of settings, often in association with other cardiac disease. Demographic and clinical factors can be utilized to profile "at-risk" patients, but the predictive value of such algorithms is low. The reasons for this presumably relate to the fact that these factors are interacting with the tissue substrate in a variable way. In addition, correlations such as these provide no insight into mechanisms associated with the development of AF in patients without other known heart disease, which is commonplace.

Over the past decade, techniques have been refined which permit an enormous amount of information relevant to disease mechanisms to be gained from examination of heart tissue. The Cardiovascular Institute has extensive experience with these techniques, and has utilized them to examine other heart disease substrates.

In this study, we propose to obtain heart tissue at the time of cardiac surgery which would otherwise be discarded. Our plan is to examine this tissue and correlate our findings with clinical data. Our hope is that the proposed study will provide insight into atrial physiology, including the molecular mechanisms underlying atrial disease and the potential development of AF.

This will be a prospective "registry" for atrial tissue. We propose an enrollment of 300 subjects, to take place at UPMC Presbyterian over a 5 year period.

Subjects will be recruited from among those patients referred for non-emergent surgery on the heart for standard indications. The patient's medical record will be reviewed and information recorded that includes demographics, heart disease history, other past medical history, current lab work, current drug therapy, and all cardiac testing the patient has undergone prior to surgery. Patients undergoing surgery will have residual atrial tissue which would otherwise be discarded (related to cannulation and/or appendectomy). Thus, obtaining this tissue will have no effect on the flow, duration, or outcome of the operative procedure.

Tissue assessment will include:

* Microscopic histology using standard tissue stains; and
* Characterization of gene expression.

Characterization of gene expression will be performed using a multiplicity of techniques which focus on DNA, RNA and proteins produced by the various cells comprising atrial tissue. Expression of a variety of genes known to be important in other cardiac diseases will be analyzed. In addition, expression of novel genes previously not known to be relevant to heart disease may be examined.

Tissue assessment data will be correlated with clinical data including preoperative AF history, demographic information, features of the medical history, details of cardiac structure/function (obtained by examining preoperative tests performed for standard indications), and the incidence of postoperative AF as a first arrhythmia diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Referred for heart surgery for standard indication
* Competent to give informed consent

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are patients of UPMC Cardiothoracic Surgery who are having standard of care CT surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schwartzman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States